CLINICAL TRIAL: NCT03435341
Title: Prospective Observational Study on Overall Survival and Quality of Life in Patients Older Than 60 Years With Acute Myeloid Leukemia Diagnosis in Spain, Treated According to Standard Clinical Practice
Brief Title: Survival in Patients Older Than 60 Years With Newly Diagnosed AML in Spain
Status: Completed | Type: Observational
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Other Study IDs: NDS-AML-001; U1111-1207-6661 (Registry Identifier: UTN)
Record Dates: First submitted 2018-02-05; First posted 2018-02-19 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-05

CONDITIONS: Leukemia, Myeloid, Acute
Keywords: Acute Myeloid Leukemia (AML); Observational; Standard Clinical Practice; Survival; Tolerability; Spain
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients diagnosed with AML: The study population will consist of approximately 150 patients over 60 with AML diagnosis according to WHO 2016 criteria.

SUMMARY:
Prospective, multicenter, observational, national study (EPA-SP) that aims to describe the survival and the quality of life, the clinical management strategies and the prognostic factors for survival related to the patient, in a prospective cohort of patients over 60 with AML diagnosis in Spain and treated outside of clinical trials; that is, under conditions of standard clinical practice.

The study will last 24 months in total from the inclusion of the first patient until the end of the last patient's follow-up

DETAILED DESCRIPTION:
Following the baseline enrolment visit, the following data corresponding to the patient's visits scheduled according to routine clinical practice will be collected in accordance with the following model:

1. Recruitment period: One year of recruitment period, data collection at the baseline visit, every 3 months in one year (month 3, 6, 9 and 12).
2. Follow-up period: data collection at the baseline visit, every 3 months in one year (month 3, 6, 9 and 12).

The patient clinical history and the study´s questionnaires will be the source documents. The study will be carried out in the facilities of the Hematology and Hemotherapy Services of the participating centers, collecting the conditions of medical action according to the standard clinical practice.

Being an observational study, no intervention out of standard clinical practice will be performed. No additional diagnostic or treatment procedures will be applied for the patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient of both sexes, aged 65 years and older.
* Any race, nationality or socioeconomic status.
* AML (defined according to WHO 2016 criteria de novo, with previous hematological history or secondary.
* Diagnosis date later than 1st November 2017 and later than each center activation date.
* Patients on first line treatment with any therapeutic strategy (intensive, attenuated or palliative).
* Having given informed consent prior to start the data collection.

Exclusion Criteria:

* Inability to understand the informed consent form.
* AML previously treated (with or without HSCT).
* Acute promyelocytic leukemia.
* Participation in a clinical trial that includes first-line treatment for AML.
* Do not grant consent.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of approximately 150 patients over 60 with AML diagnosis, defined according to World Health Organization (WHO) 2016 criteria (presence of blasts in the bone marrow or peripheral blood equal to or greater than 20%).
  Due to the observational and descriptive nature of the present investigation, the inclusion of a control group is not considered.
Sampling Method: Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2018-02-28 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
The median survival time in adult patients over 60 with AML diagnosis | Up to approximately 12 months
  The overall survival will be calculated, defined as the time from the diagnosis date to the death date from any reason. In patients who have not died (censored) at the time of data collection, it will be considered the available time to the last control (or last date). The overall survival will be analyzed using the Kaplan-Meier method, providing the median at 95% CI. Patients who undergo a hematopoietic transplant will be censored at that time.

SECONDARY OUTCOMES:
Overall Survival | Up to approximately 12 months
  The Kaplan Meier curve, with the median and the lower and upper limits of the 95% confidence interval, will be reported.
To describe the socio-demographic and clinical characteristics of patients | Up to approximately 12 months
  A description of the study socio-demographic and clinical variables will be made. The distributions of absolute and relative frequencies of the qualitative variables will be reported, as well as the measures of central and dispersion tendency of the quantitative variables. A 95% CIs will be obtained for the main variables.
To describe the disease characteristics | Up to approximately 12 months
  A description of the variables that characterize the disease under study will be made. The distributions of absolute and relative frequencies of the qualitative variables will be reported, as the measures of central tendency and dispersion of the quantitative variables. A 95% CIs will be obtained for the main variables.
To describe the front-line treatment strategies | Up to approximately 12 months
  The frequency distributions for the first lines of treatment will be presented, as well as the rate distribution of the most frequent treatment sequences and their evolution. It will be reported the descriptive statistics period of the first treatment lines.
To assess the HRQOL evolution over time | Up to approximately 12 months
  Descriptive statistics will be reported for each of the five dimensions at every period of application of the EQ-5D, so as an overall lineal model of repeated measures for the VAS.
To evaluate the impact on early mortality | Up to approximately 8 weeks
  The t-test will be used to evaluate the impact of the initial leukocyte count on early mortality (dichotomous variable minus death or not in the first 8 weeks). The stratified analysis with the same approach will be done for treatments that achieve a sufficient sample.
To evaluate the prognostic impact on overall survival | Up to approximately 12 months
  A Cox regression model will be made considering the patient survival as a dependent variable and as possible factors the subjective variables (asthenia and HRQOL) at the time of diagnosis, the patient's general condition, and any other clinical variable that is evaluated as possible predictor. No more than 10 independent variables will be included in the model for theoretical reasons.
To explore the scales scores to be used as potential predictors tools of treatment tolerability in patients with newly diagnosed AML. | Up to approximately 12 months
  The therapeutic approach will be collected according to the investigator clinical judgment, the score of each of the items on the Lee and GAH scales and the treatment administered tolerability assessment according to the score obtained in each scale. The weighting coefficients will be calculated using a complete multiple linear regression model and a multiple logistic regression. The optimal cut points for use as a predictive tool for treatment tolerability will be determined by using the ROC curve technique.

CONTACTS AND LOCATIONS:
Overall Officials: Montserrat Rafel, RML Advocacy, Study Director — Celgene
Locations (40):
- Spain (40):
  - Hospital de Jerez, Jerez de la Frontera, Andalucía/Cádiz
  - Hospital Virgen de las Nieves, Granada, Andalucía/Granada
  - Hospital Carlos Haya, Málaga, Andalucía/Málaga
  - Hospital Virgen del Rocio, Seville, Andalucía/Sevilla
  - Hospital Universitario Nuestra Señora de Valme, Seville, Andalucía/Sevilla
  - Hospital Univ. Reina Sofia, Córdoba, Andalusia
  - Hospital Universitario Virgen Macarena, Seville, Andalusia
  - Hospital Clínico Lozano Blesa, Zaragoza, Aragon
  - Hospital Son Espases, Palma de Mallorca, Balearic Islands
  - Hospital de Basurto, Bilbao, Vizcaya, Basque Country
  - Hospital Universitario de Donostia, San Sebastián, Guipúzcoa, Basque Country
  - Hospital de Txagorritxu, Vitoria-Gasteiz, Basque Country
  - Hospital Dr. Negrín, Las Palmas de Gran Canaria, Canary Islands
  - Hospital Nuestra Señora de Candelaria, Santa Cruz de Tenerife, Canary Islands
  - Hospital Universitario Canarias, Santa Cruz de Tenerife, Canary Islands
  - Hospital Universitario de Burgos, Burgos, Castille and León
  - Hospital de León, León, Castille and León
  - Complejo Hospitalario de Salamanca, Salamanca, Castille and León
  - Clínico de Valladolid, Valladolid, Castille and León
  - Hospital del Mar, Barcelona, Catalonia
  - Hospital Arnau de Vilanova Lleida, Lleida, Catalonia
  - Hospital de Althaia (H. Sant Juan de Deu de Manresa), Manresa, Barcelona, Catalonia
  - Hospital Infanta leonor, Madrid, Comunidad Madrid
  - Hospital Infanta Cristina, Badajoz, Extremadura
  - Complejo Hospitalario Universitario de A Coruña, A Coruña, Galicia
  - Complejo Hospitalario Universitario de Orense, Ourense, Galicia
  - Hospital Santa Lucía, Cartagena, Murcia, Murcia
  - Complejo Hospitalario de Navarra, Pamplona, Navarra, Navarre
  - Hospital Universitario Cabueñes, Gijón, Principality of Asturias
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital General Alicante, Alicante, Valencia
  - Hospital General Universitario de Valencia, Valencia, Valencia
  - Hospital Universitario La Princesa, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Fundación Jiménez Díaz, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital de Fuenlabrada, Madrid
  - Hospital de Getafe, Madrid